CLINICAL TRIAL: NCT00238966
Title: A One Arm, Open-label Study to Investigate the Tolerability and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in Renal Transplant Recipients Who Received Mycophenolate Mofetil (MMF)
Brief Title: Extension Study to Assess Tolerability and Safety of Enteric-coated Mycophenolate Sodium in Renal Transplant Recipients Who Received Mycophenolate Mofetil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405DE02E1
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
This extension study is considered to allow patients being treated with EC-MPS to collect further information on the long-term safety of this drug.

ELIGIBILITY:
Inclusion/ Exclusion criteria

- Only patients who were participating in study CERL080A2405-DE02 and have completed the first 6 months of the core study can be included in this additional extension study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2002-11; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability based on adverse events within 6 months after switching patients from MMF to optimized enteric-coated mycophenolate sodium.

SECONDARY OUTCOMES:
Safety based on renal function within 6 months after medication switch.
Pharmacokinetics (PK) in a randomized subpopulation.
Efficacy measured by the incidence of biopsy-proven acute rejection, graft loss or death within 6 months post medication switch.
Efficacy measured by the incidence of biopsy-proven acute rejection 6 months post medication switch.
Graft survival and patient survival 6 months post medication switch.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis